CLINICAL TRIAL: NCT00046150
Title: 12-Week, Multinational, Multicenter, Controlled, Open, 1:1 Randomized, Parallel Clinical Trial Comparing the Safety of HMR1964 and Insulin Aspart Used in Continuous Subcutaneous Insulin Infusion (CSII) in Subjects With Type 1 Diabetes Mellitus
Brief Title: 12 Week,Comparing Safety of HMR1964 & Insulin Aspart Used in Continuous Subcutaneous Infusion in Type 1 Diabetes.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMR1964/3006; HMR1964
Record Dates: First submitted 2002-09-20; First posted 2002-09-23 (Estimated); Last update posted 2008-06-19 (Estimated); Status verified 2008-06

CONDITIONS: Diabetes, Type I
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — insulin glulisine

INTERVENTIONS:
Drug: Insulin glulisine (HMR1964)

SUMMARY:
The purpose of this study is to compare the safety of HMR 1964 and insulin aspart when used in external pumps with respect to catheter occlusions, GHb assessment, insulin doses, blood glucose parameters, hypoglycemic episodes, unexplained hyperglycemia, adverse events, laboratory data, and vital signs.

ELIGIBILITY:
INCLUSION CRITERIA:

Subjects meeting all of the following criteria will be considered for enrollment into the study:

* Men and women above the age of 18.
* Women are either not of childbearing potential (surgically sterile, or postmenopausal for more than 2 years) or are not pregnant and agree to use a reliable contraceptive measure for the duration of the study. Reliable contraceptive measures include the follows: systemic contraceptive (oral, implant, injections), diaphragm with intravaginal spermicide, cervical cap, intrauterine device, or condom with spermicide.
* Type 1 diabetes mellitus as established in the medical history (for the purpose of this protocol: onset of diabetes under the age of 40 and has required continuous insulin therapy since diagnosis).
* At least 1 year of continuous insulin treatment with at least 6 months of continuous subcutaneous insulin infusion treatment immediately prior to study entry.
* Use of the same type of external insulin pump (MiniMed programmable pump, or Disetronic pump type H Tron Plus V 100 or D Tron) for at least 3 months prior to study entry.
* HbA1c <8.5% measured at visit 1.
* Ability and willingness to perform blood glucose monitoring using the sponsor-provided blood glucose meter and subject diary at home.

Informed consent must be obtained in writing for all subjects at enrollment into the study (see Section 12.3).

EXCLUSION CRITERIA:

Subjects presenting with any of the following will not be included in the study:

* Active proliferative diabetic retinopathy, as defined by the application of focal or panretinal photocoagulation or vitrectomy, in the 6 months prior to visit 1, or any other unstable (rapidly progressing) retinopathy that may require surgical treatment (including laser photocoagulation) during the study.
* Diabetes other than type 1 diabetes mellitus.
* History of serious ketosis episode requiring hospitalization in the 3 previous months.
* History of abscess at the infusion site in the previous 3 months.
* Pancreatectomised subjects.
* Subjects who have undergone pancreas and or islet cell transplants.
* Likelihood of requiring treatment during the study period with drugs not permitted by the study protocol (see Section 6.2).
* Treatment with any investigational drug in the last month before visit 1.
* History of seizure disorders.
* History of hypersensitivity to insulin or insulin analogues or any other excipients in the HMR1964 or insulin aspart formulation (see the Global Investigators Brochure [7] and the insulin aspart SPC [13] for a list of excipients).
* Clinically relevant cardiovascular, hepatic, neurologic, endocrine, active cancer, or other major systemic disease making implementation of the protocol or interpretation of the study results difficult or would, in the opinion of the investigator, preclude the safe participation of the subject in this protocol.
* History of drug or alcohol abuse.
* Impaired hepatic function, as shown by but not limited to ALT or AST greater than twice the normal upper limit measured at visit 1.
* Impaired renal function, as shown by but not limited to serum creatinine >177 micromol/L (>2.0 mg/dL) measured at visit 1.
* Pregnancy (as determined by pregnancy blood test at visit 1) or breast-feeding.
* Night shift workers.
* Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.
* Subject unlikely to comply with protocol, e.g. an inability and unwillingness to participate in adequate training, an uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study.
* Employee of the sponsor or of sponsor representatives.
* Subjects who have previously been treated with HMR1964.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2002-05; Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Frequency of catheter occlusions

SECONDARY OUTCOMES:
Unexplained hyperglycemia, parameters of glycemic control

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (3):
- Hospital de Rangueil, Toulouse, France
- Sanofi-aventis Administrative Office, Berlin, Germany
- Sanofi-aventis Administrative Office, Gouda, Netherlands

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com